CLINICAL TRIAL: NCT06921694
Title: A Combined Exercise Programme Involving Strengthening, Flexibility and Aerobic Exercise for Lower Back Pain: a Randomised-controlled Study
Brief Title: A Combined Exercise Programme Involving Strengthening, Flexibility and Aerobic Exercise for Lower Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Kimberley Edwards, Professor Sport Exercise and Nutrition Education, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMHS 279 0423
Record Dates: First submitted 2025-03-26; First posted 2025-04-10 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-04

CONDITIONS: Low Back Pain, Chronic
Keywords: chronic non specific low back pain; exercise intervention
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Masking Description: It is not possible to blind/mask the investigators or participants due to the nature of the intervention (i.e. they know what exercise they are doing). However a different person undertakes the randomisation to keep that separate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Participants continue with their usual exercise regime.
- Runner Group (Experimental): Particpants follow an 8 week intervention including aerobic elements (running), a schedule of gradually intensitfing strengthening exercises and flexibility exercises.
  Interventions: Behavioral: Runner group
- Swim/Cycle group (Experimental): Particpants follow an 8 week intervention including aerobic elements (swim/cycle), a schedule of gradually intensitfing strengthening exercises and flexibility exercises.
  Interventions: Behavioral: Swim/Cycle Group

INTERVENTIONS:
Behavioral: Runner group — The intervention groups undertake 8 weeks of a combined exercise programme including aerobic elements (running), a schedule of gradually intensifying strengthening exercises and flexibility exercises
  Arms: Runner Group
Behavioral: Swim/Cycle Group — The intervention groups undertake 8 weeks of a combined exercise programme including aerobic elements (swim/cycle), a schedule of gradually intensitfing strengthening exercises and flexibility exercises
  Arms: Swim/Cycle group

SUMMARY:
This randomised controlled trial will evaluate the effectiveness of different exercise modalities for individuals with low back pain. Participants will be allocated to one of three groups: a control arm (usual exercise), a running-based intervention, or a swimming/cycling-based intervention. Outcomes related to pain and function will be measured at baseline, 8 weeks, and 12 months.

DETAILED DESCRIPTION:
This study is designed to assess the impact of structured exercise interventions on pain and functional outcomes in otherwise healthy adults with low back pain. Eligible participants recruited from the community will be randomised into one of three arms: (1) control group, continuing their usual exercise activities; (2) running intervention group; or (3) swimming/cycling intervention group.

The two intervention arms will complete an 8-week combined exercise programme consisting of aerobic training (running or swimming/cycling, depending on group assignment), progressive resistance training, and prescribed flexibility exercises. The programme is structured to gradually increase in intensity over the 8-week period to enhance adherence and minimize risk of injury.

Efficacy will be evaluated using validated patient-reported outcome measures (PROMs) capturing pain intensity and functional capacity. These assessments will be administered at three time points: baseline (prior to the intervention), post-intervention (8 weeks), and long-term follow-up (12 months). This design will enable analysis of both the short-term and sustained effects of exercise modality on low back pain management.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45 years
* Participant is willing and able to give informed consent for participation in the study
* Suffering from chronic NSLBP (more than 3 months, localised below the costal margin and above the gluteal folds)
* Suffers from pain or functional limitations as a result of their LBP (minimum VAS (back) score of 3/10 or ODI score of at least 5/50 or RMD score of at least 5/24 (note, unlike ODI, RMD does not describe specific cuts offs for different levels of disability)
* Able to exercise

Exclusion Criteria:

* Radiating pain to leg / sciatica / acute radiculopathy
* Specific diagnosis/condition for LBP (e.g. herniated disk, degenerative disk disease, spondylolysis, spinal stenosis, spinal tumour, facet joint damage)
* History of osteoporosis , arthritis, scoliosis, or kyphosis.
* Current spinal infection, cancer or a current fracture (any bone).
* History of spinal/back surgery
* Unable to participate in physical activity and exercise
* Pregnant or breast feeding
* History of substance abuse
* History of psychiatric illness (eg. depression, dementia, schizophrenia) for which currently taking medication
* History or current neurological condition (e.g. epilepsy)
* Not in possession or have access to adapted equipment (phone, computer, functioning WIFI)
* Unable to understand and communicate in English
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
VAS pain score | Baseline, 8 weeks, 12 months
  VAS pain score on 100 point scale
  * Range: 0 to 100
  * Anchors: 0 = no pain, 100 = worst imaginable pain
  * Interpretation: Higher scores indicate worse pain

SECONDARY OUTCOMES:
Oswestry disability index | Baseline, 8 weeks, 12 months
  Oswestry disability index (PROM questionnaire)
  * Range: 0 to 100 (expressed as a percentage)
  * Anchors: 0 = no disability, 100 = maximum disability
  * Interpretation: Higher scores indicate greater disability
Roland Morris Disability questionnaire | Baseline, 8 weeks, 12 months
  Roland Morris Disability questionnaire (PROM questionnaire)
  * Range: 0 to 24 (some versions extend to 0-23 or 0-25 depending on adaptation, but 0-24 is most common)
  * Anchors: 0 = no disability, 24 = maximum disability
  * Interpretation: Higher scores indicate greater disability

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley Edwards, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Queen's Medical Centre, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
This is a small study with limited administrative support.